CLINICAL TRIAL: NCT01356459
Title: A Prospective Randomised Controlled Trial of the Effectiveness of Absorbent Silicone Self Adherent Dressings in the Prevention of Sacral and Heel Pressure Ulcers in Trauma and Critically Ill ED/ICU Patients
Brief Title: Pressure Ulcer Prevention in Intensive Care Unit (ICU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010.261
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Pressure Ulcers
Keywords: Pressure ulcers; ICU; Prevention
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Patients in this arm will have Mepilex dressings applied to their sacrum and heels
  Interventions: Device: Mepilex Border Dressing
- Control (No Intervention): Patients in this arm will have standard care

INTERVENTIONS:
Device: Mepilex Border Dressing — Soft silicone self adherent dressing
  Other Names: Mepilex Border Sacrum; Mepilex Heel
  Arms: Intervention

SUMMARY:
The study is designed as a randomised controlled trial of trauma patients admitted to the Royal Melbourne Hospital (RMH) Emergency Department (ED) and subsequently transferred to the Intensive Care Unit (ICU). Patients meeting the study inclusion criteria will be randomly allocated to either the control group that will receive usual pressure ulcer prevention strategies or the trial group that will receive usual care plus have a Mepilex Border Sacrum dressing applied to their sacrum and Mepilex Boarder Heel dressing applied to each heel in the ED.

Hypothesis:Patients treated with Mepilex Border dressings will have a lower incidence rate of sacral and heel pressure ulcer development than patients receiving standard care.

DETAILED DESCRIPTION:
Aims

To determine the effectiveness of Mepilex Border dressings in preventing sacral and heel pressure ulcer development

To determine the cost effectiveness of Mepilex Border dressings in preventing sacral and heel pressure ulcers.

Primary endpoint

Incidence rates of pressure ulcers in ICU expressed as the total number of pressure ulcers developed per week in both groups

Secondary endpoint

Cost of trial dressings to prevent pressure ulcers Cost of the management of developed pressure ulcers

Hypothesis

Patients treated with Mepilex Border dressings will have a lower incidence rate of sacral and heel pressure ulcer development than patients receiving standard care.

Subjects and Sampling

All trauma and critically ill patients admitted to ED and defined by the ED as being trauma and/or critically ill. These patients will subsequently be transferred to ICU over a six (6) month period commencing January 2010

Sample size

The investigators calculate that to detect a decrease in the ICU pressure ulcer incidence rate of 3.5% (from 4% to 0.5%) in the intervention group with power set at 80% and alpha of 0.05 will require a total of 220 patients per group.

Randomisation

Subjects will be randomised to either the intervention group or to the control group by allocating each subject a study number and then using a computer generated set of random numbers to determine group allocation. The randomisation of participants will be undertaken by an ED research nurse when the patient is admitted to ED and following screening to determine if they meet the inclusion criteria.

Participant selection:

The following procedure will be used by the ED Research Nurse to determine if the person is included in the study and to which group the individual will be allocated.

Potential participant Meets inclusion criteria and does not meet exclusion criteria Conducts standard MH pressure ulcer risk screening (Braden Scale) Assigns participant a study number Records ED data at admission (see below) Determines group allocation by comparing participant study number to randomisation sequence

If randomised to trial group:

Applies Mepilex Border dressings to sacrum and heels Records time of dressing application

Intervention

Trial group patients who meet the inclusion criteria will have a Mepilex Border dressing applied to their sacrum and heels on admission to ED by the ED research nursing staff. It is necessary to apply the dressing at this point because the investigators wish to investigate the potential protective effects of the dressing if the patient needs to have a surgical procedure which may involve a long period in the OR.

Mepilex Border Dressing Mepilex Border is an absorbent, atraumatic self-adhesive island dressing with a perforated soft silicone wound contact layer. The absorbent core of the dressing consists of three components, a thin sheet of polyurethane foam, a piece of nonwoven fabric and a layer of superabsorbent polyacrylate fibres. The core is located centrally upon a larger piece of polyurethane film and is held in place by the perforated silicone adhesive layer that extends to the outer margins of the dressing. This gentle adhesion also tends to prevent maceration by inhibiting the lateral movement of exudate from the wound on to the surrounding skin. The silicone layer does not adhere to the surface of a wound and therefore the dressing may be removed without causing pain or trauma.

Method of use The wound contact surface of the dressing is protected with a divided plastic film, which must be removed before use. If clinically indicated, the wound should be cleaned and the surrounding skin thoroughly dried before application of the dressings. If additional fixation is required this should only be applied around the margins of the dressing.

Frequency of Change The interval between changes will normally be determined by the amount of exudate produced by the wound, but the dressing may be left in place for several days on clean non-infected wounds.

The manufacturers note that there are no absolute contra-indications to the use Mepilex Border dressings.

As patients in this study will not have a wound in the areas where the dressing will be applied the investigators propose to change each dressing every three days or as required if they become soiled or dislodged. This decision will be made by members of the research team whao are involved with the daily assessment of each patient.

The skin under the dressings will be observed daily by members of the research team to determine if any pressure related injuries have developed. Pressure related injuries are defined as per the Australian Wound management Association clinical guideline for the prediction, prevention and management of pressure ulcers. All members of the research team have undergone inter-rater reliability testing in September 2010 for their ability to recognise and stage a pressure ulcer.

Measurement

Patient demographics Age Wt Gender Race Pre-existing disease Charlson Comorbidity Index score Reason for admission Management pre admission Eg. Time on spinal board Time in Ambulance Time in ED ED management - ventilation ED physiological observations Number of OR procedures Time in OR Time in ICU Nutritional status Immobility Urinary incontinence Faecal incontinence

Pressure ulcers:

Pressure ulcer incidence per week

Pressure ulcers will be staged according to the Australian Wound Management Association (AWMA) staging system

Cost of trial dressings used for total duration of trial Cost of management of developed pressure ulcers Staff time Consumables

Physiological data All physiological data collected in ICU Shock/SIRS Cardiac arrest Drive lines Spinal cord injury Mechanical ventilation Traction/external fixators

Pharmaceutical data All drugs Sedation/Paralytics Vasopressor drugs

Analysis

A survival analysis will be used to determine the difference in pressure ulcer incidence rates per group and logistic regression will be used to investigate potential interactions between demographic and physiological variables between groups and incidence rates. Analysis will be conducted separately for sacral and heel wounds as the main analysis. The investigators may pool the results if there appears to be no difference between the incidence rates for sacral and heel wounds. All analytical procedures will be carried out by the Statistical Consulting Centre, University of Melbourne.

Cost analysis will involve calculating the total treatment and prevention costs associated with pressure ulcers including staff time and consumables. The costing analysis will be carried out by a research nurse in ICU who will observe and record the total staff time by grade of RN spent on pressure ulcer prevention in all patients. Costs such as support surfaces (dynamic mattresses and overlays) will also be added to prevention costs. Intervention group patients will also have the costs of the Mepilex Border dressings added to their pressure ulcer prevention costs.

Should a patient in either group develop a pressure ulcer the cost of managing the wound will be calculated based on staff time by grade, consumables such as dressings, investigations such as microbiological specimen collection and analysis. These costs will be determined for the total time that the patient remains in ICU.

ELIGIBILITY:
Inclusion Criteria:

* ED and ICU admission for critical illness and/or major trauma Over 18 years old

Exclusion Criteria:

* Less than 18 years old Suspected or actual spinal injury Pre-existing sacral or heel pressure ulcer Trauma to sacral and/or heel area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Pressure ulcer incidence | Weekly
  Number of pressure ulcers developed in the ICU per week

SECONDARY OUTCOMES:
Cost | Weekly
  The cost of treating developed pressure versus the cost of preventing the development of pressure ulcers

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Melbourne Hospital, Melbourne, Victoria, Australia